CLINICAL TRIAL: NCT04873271
Title: Evaluation of Implantable Tibial Neuromodulation (TITAN 1) Feasibility Study
Acronym: TITAN 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT20033
Record Dates: First submitted 2021-04-28; First posted 2021-05-05 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Neoplasm Staging; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Medtronic Implantable Tibial Neuromodulation (TNM) System — Tibial neuromodulation (TNM) devices are implantable devices that provide stimulation to the tibial nerve.

SUMMARY:
This is a prospective, multicenter, feasibility study to characterize the procedure for the implantable TNM device in subjects with overactive bladder.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Primary Inclusion Criteria:

1. Subjects 18 years of age or older
2. Have a diagnosis for at least 6 months of OAB
3. No OAB pharmacotherapy for 2 weeks prior to the baseline voiding diary
4. Willing and able to accurately complete study diaries, questionnaires, attend visits, operate the system and comply with the study protocol
5. Willing and able to provide signed and dated informed consent

Primary Exclusion Criteria:

1. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury
2. Severe uncontrolled diabetes
3. History of urinary retention within the previous 6 months
4. Current symptomatic urinary tract infection
5. Have primary stress incontinence or mixed incontinence where the stress component overrides the urge component
6. Current urinary tract mechanical obstruction
7. Have knowledge of planned magnetic resonance imaging (MRIs) or diathermy
8. History of a prior implantable tibial neuromodulation system
9. Skin lesions or compromised skin integrity at the implant site
10. Anatomical defects, clinically significant edema or previous surgeries which precludes use of the device
11. Previous pelvic floor surgery in the last 6 months
12. Women who are pregnant or planning to become pregnant
13. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements.
14. Any subject who is considered to be part of a vulnerable patient population.
15. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results.** **Subjects in concurrent studies can only be enrolled with permission from Medtronic.

Contact Medtronic's study manager to determine if the subject can be enrolled in both studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
To characterize the TNM device implant procedure | 14 days
  This information will be collected through a series of questions for participating investigators via a case report form at implant through the 14-day follow-up visit.
To characterize the TNM device initial system use | 14 days
  This information will be collected through programming and device data at implant through the 14-day follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Miller, Study Director — Medtronic
Locations (7):
- United States (7):
  - Georgia Urology, Marietta, Georgia
  - Urologic Research and Consulting, Englewood, New Jersey
  - FirstHealth Urogynecology, Hamlet, North Carolina
  - Prisma Health, Greenville, South Carolina
  - Sanford Health, Sioux Falls, South Dakota
  - Urology Partners of North Texas, Arlington, Texas
  - Milwaukee Urogynecology Ascension Medical Group, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No